CLINICAL TRIAL: NCT03291678
Title: Randomized Control Study for Patient With Abdominal Undescended Testis Using New Technique
Brief Title: Impact of Percutaneous Laparoscopic Assisted Internal Ring Ligation During Lap Orchiopexy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ahmed Hamdy Rateb (Other)
Collaborators: Assiut University (Other)
Responsible Party: Sponsor-Investigator, Ahmed Hamdy Rateb, resident physician of general surgery assuit university, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASSUIT HOSPITAL UNIVERSITY
Record Dates: First submitted 2017-09-08; First posted 2017-09-25 (Actual); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Congenital Disorders
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities

STUDY DESIGN:
Intervention Model Description: one group which is control group will not subjected to internal ring ligation and another group will subjected to closure of the internal ring
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- new laparoscopic orchiopexy (Experimental): this group will subjected to classic laparoscopic orchiopexy by delivery of abdominal undescended testis to subdartos pouch of scrotum with closure of internal ring
  Interventions: Procedure: new laparoscopic orchiopexy
- classic laparoscopic orchoipexy (Active Comparator): this group will subjected to classic laparoscopic orchiopexy by delivery of abdominal undescended testis to subdartos pouch of scrotum
  Interventions: Procedure: classic laparoscopic orchiopexy

INTERVENTIONS:
Procedure: new laparoscopic orchiopexy — closure of the internal ring of the inguinal canal after descending of the testis to scrotum using needle percutaneous
  Arms: new laparoscopic orchiopexy
Procedure: classic laparoscopic orchiopexy — delivery of abdominal testis into scrotum without closure of the internal ring of the inguinal canal
  Arms: classic laparoscopic orchoipexy

SUMMARY:
Impact of percutaneous internal ring ligation during laparoscopic orchiopexy in decreasing incidence of congenital hernia

DETAILED DESCRIPTION:
Cryptorchidism is the most common genitourinary anomaly in male children. Its incidence can reach 3% in full term neonates, rising to 30% in premature boys . The treatment of the crypt orchid testicle is justified by the increased risk of infertility and malignancy, as well as an associated inguinal hernia and the risk of trauma to the ectopic testicle against the pubis. Furthermore, the psychological stigma of a missing testis for the patient, as well as the parents' anxiety is also factors that justify this type of treatment .

About 20% of crypt orchid testicles are non palpable. The treatment of non-descended testicles is mandatory due to the increased risk of infertility, present in up to 40% of the patients, as compared to 6% of control groups, including malignancy, which reaches 20 times that of normal adults .

The treatment of the crypt orchid testis before 2 years of age is recommended, treatment is necessary not only for the risk of malignancy, but also for the satisfaction and improvement in the quality of the patient's life and parents´ concern for their children's health.

In relation to diagnosis, despite a sensitivity of 70-90% in the diagnosis of inguinal testes, ultrasonography is not useful in intra-abdominal cases . Although presenting a better quality, both computed tomography and nuclear magnetic resonance lack sufficient sensitivity and specificity to be considered as gold standard diagnostic tools . More recently, the magnetic angioresonance was introduced with sensibility of 96% and specificity of 100%, but it is still a new method, with high costs, also requiring general anesthesia in children .

In relation to the treatment, the use of gonadotrophin for un descended testes presents a success rate of definitive descent to the scrotum of 21 to 56%, with better results in bilateral cases . Surgical treatment via an inguinal incision is the main treatment option for palpable testicles, but can also be employed for the evaluation and treatment of non-palpable testis. In this situation, however, surgical exploration can often require large incisions and extensive dissections, especially in bilateral cases. This can be avoided using laparoscopic evaluation, with a sensitivity and specificity reaching more than 90%

ELIGIBILITY:
* INCLUSION CRITERIA

  1. Age above six months
  2. SEX must be male
  3. Surgical approach is closure of internal ring via percutaneous technique after delivery of undescended testis
* EXCLUSION CRITERIA

  1. Age less than 3 months
  2. Patients with palpable undescended testis
  3. Any associated major congenital anomalies like cardiac anomalies

Ages: 6 Months to 2 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2017-09-25 (Estimated); Primary Completion 2018-09-05 (Estimated); Study Completion 2018-09-06 (Estimated)

PRIMARY OUTCOMES:
decrease incidence of congenital hernia which associated with undescended testis | one year
  patient follow up will be after 15 days and then after two months by examination of the operation site ,stitches , and hernial orifices to be sure of absence of congenital hernia

SECONDARY OUTCOMES:
The secondary outcome measure postoperative complication | one week post operative
  close observation of the patient depending on follow up the wound daily ,occurence of edema by observation, good feeding of the patient by mother

CONTACTS AND LOCATIONS:
Overall Officials: gamal abdel hamid ahmed, prof, Principal Investigator — prof of general surgery assuit university

IPD SHARING:
Plan to Share IPD: Undecided